CLINICAL TRIAL: NCT00278967
Title: An Efficacy Evaluation of 2 Different Bowel Cleansing Preparations in Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F38-26
Record Dates: First submitted 2006-01-13; First posted 2006-01-19 (Estimated); Last update posted 2006-10-19 (Estimated); Status verified 2006-10

CONDITIONS: Colonoscopy
Keywords: colonoscopy; preparation
MeSH Terms: interventions — Bisacodyl

INTERVENTIONS:
Drug: HalfLytely with Bisacodyl Tablets Bowel Prep Kit
Drug: HalfLytely - Reformulation

SUMMARY:
To compare the safety and efficacy of 2 different bowel cleansing preparations prior to colonoscopy in adult subjects.

DETAILED DESCRIPTION:
The goal of the study is to evaluate the efficacy of 2 different HalfLytely preparations to produce a clinically acceptable degree of cleansing of the bowel, sufficient for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

- Male or female outpatients who are undergoing colonoscopy for the following routinely accepted indications:

Evaluation of BE results GI bleeding Anemia of unknown etiology Neoplastic disease surveillance Endosonography Inflammatory bowel disease Unknown diarrhea or constipation etiology Polypectomy Laser therapy Routine Screening

* At least 18 years of age
* Otherwise in good health, as determined by physical exam and medical history
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, sterilized, abstinent, or vasectomized spouse)
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, or toxic megacolon
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration
* Subjects who are undergoing colonoscopy for foreign body removal and decompression
* Subjects with pre-existing electrolyte disturbances, such as dehydration, or those secondary to the use of diuretics
* Subjects who are taking drugs that may affect electrolyte levels
* Subjects taking laxatives or prokinetic agents that refuse to discontinue these treatments for the duration of the study
* Subjects with known clinically significant electrolyte abnormalities such as hypernatremia, hyperphosphatemia, hypokalemia, or hypocalcemia
* Subjects who are pregnant or lactating, or intending to become pregnant during the study
* Subjects of childbearing potential who refuse a pregnancy test
* Subjects who are allergic to any preparation components
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2006-02; Study Completion 2006-08

PRIMARY OUTCOMES:
Efficacy - preparation quality using a 4-point scale

SECONDARY OUTCOMES:
Safety - patient-reported preparation related side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, M.D., Principal Investigator — Long Island GI Research Group
Locations (10):
- United States (10):
  - Anaheim, California
  - Jupiter, Florida
  - Miami, Florida
  - Baton Rouge, Louisiana
  - Laurel, Maryland
  - Great Neck, New York
  - Raleigh, North Carolina
  - Germantown, Tennessee
  - Bellevue, Washington
  - Spokane, Washington